CLINICAL TRIAL: NCT06021795
Title: Sounds for Sleep Study in Patients Suffering From Moderate to Severe Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Wave Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-006
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Treatment using a customized sound audio track delivered via standard commercially available bone conduction headsets
  Interventions: Device: Sound Treatment

INTERVENTIONS:
Device: Sound Treatment — Customized sound audio track delivered via standard commercially available bone conduction headset

SUMMARY:
Assess the effect of a customized audio track delivered via standard commercially-available bone conduction headsets on the quality of sleep

DETAILED DESCRIPTION:
A single-center study in 25 subjects suffering from moderate to severe insomnia and assess the effectiveness of the intervention. Intervention consists of treatment using a customized audio track delivered via standard commercially-available bone conduction headsets daily for four (4) weeks. Effectiveness is defined by a statistically significant improvement in Insomnia Severity Index (ISI) and Pittsburgh Sleep Quality Index (PSQI) at baseline versus the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Meets DSM 5 criteria for insomnia disorder
* Insomnia Severity Index (ISI) of 15 - 28

Exclusion Criteria:

* Use of sleep medications, sedating or alerting medications or antidepressants in the last 3 months
* Diagnosis of any autoimmune disorder or any medical or sleep disorder that could affect sleep
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | 4 weeks
  Reduction in Insomnia Severity

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  Reduction in Sleep Quality

CONTACTS AND LOCATIONS:
Overall Officials: Elan Hekier, MD, Principal Investigator — San Francisco Otolaryngology Medical Group
Locations (1):
- San Francisco Otolaryngology Medical Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No